CLINICAL TRIAL: NCT05672459
Title: A Phase 1/2a, Safety And Efficacy Study Of HLA-G- Targeted CAR-T Cells IVS-3001 In Subjects With Previously Treated Advanced HLA-G-Positive Solid Tumors
Brief Title: A Safety And Efficacy Study Of HLA-G- Targeted CAR-T Cells IVS-3001 In Subjects With Previously Treated Advanced HLA-G-Positive Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Invectys (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0261; NCI-2023-00020 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: IVS-3001; CART; HLA-G; ccRCC-renal cell carcinoma; Kidney cancer; EOC-epithelial ovarian cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — fludarabine phosphate; Cyclophosphamide; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Part 1) and Expansion (Part 2 ) (Experimental): Participants will receive IVS 3001 at the selected dose Participants will receive IVS 3001 at the recommended phase 2 dose
  Interventions: Drug: Single Injection of IVS-3001- Anti - HLA-G CAR-T cells; Drug: Fludarabine phosphate; Drug: Cyclophosphamide; Procedure: leukapheresis

INTERVENTIONS:
Drug: Single Injection of IVS-3001- Anti - HLA-G CAR-T cells — Given by IV (vein)
Drug: Fludarabine phosphate — Given by IV (vein)
Drug: Cyclophosphamide — Given by IV (vein)
Procedure: leukapheresis — Given by IV (vein)

SUMMARY:
The proposed clinical study is a Phase 1/2a trial to investigate the safety, tolerability, pharmacokinetics and clinical activity of anti-HLA-G CAR-T cells IVS-3001 administered to subjects with previously treated, locally advanced, or metastatic solid tumors which are HLA-G positive (HLA-G+) - as determined by immunohistochemistry (IHC) analysis on tumor biopsies using the 4H84 antibody.

DETAILED DESCRIPTION:
Primary Objectives:

IVS-3001 is an autologous CAR-T cell therapy targeting human leukocyte antigen (HLA-G)

* Phase 1: To determine the safety, tolerability and the recommended phase 2 dose (RP2D) of IVS-3001 in subjects with refractory or relapsed HLA-G+ solid tumors.
* Phase 2a: To evaluate the anti-tumor activity of IVS-3001 in selected HLA-G+ solid tumor types.

Secondary Objectives:

* To evaluate pharmacokinetic profile of IVS-3001: persistence, expansion.
* To evaluate the clinical activity of IVS-3001 in selected HLA-G+ solid tumor types.
* To assess the long-term safety of IVS-3001.

Exploratory Objectives:

• To explore functionality of IVS-3001 as well as immune biomarkers linked with IVS-3001 and their relationship with clinical response

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Histologically or pathologically confirmed diagnosis of a locally advanced unresectable or metastatic HLA-G+ select solid tumor malignancy who failed or intolerant to standard of care therapies known to confer clinical benefit per treating physician.

   For Phase 2a, eligible subjects will be enrolled into indication-specific cohorts:
   1. Cohort 1: HLA-G+ clear cell renal cell carcinoma who failed or intolerant to checkpoint inhibitor (CPI) and tyrosine kinase inhibitor (TKI)
   2. Cohort 2: Epithelial ovarian carcinoma who failed or intolerant to platinum-based therapy, and should have failed or intolerant for PARP inhibitor if BRCA 1/2 mutated
   3. Cohort 3: Other HLA-G+ tumors (biomarker driven) who failed or intolerant to at least one prior line of therapy and for whom at discretion of treating physician there is no standard therapy to confer a clinical benefit
3. HLA-G expression on tumor cells (any level of expression is acceptable) as determined by immunohistochemistry (IHC) analysis on tumor biopsies using the 4H84 antibody [1, 2]
4. Measurable disease (at least one target lesion) per RECIST v1.1 [3]
5. Life expectancy >12 weeks.
6. Availability of a pre-treatment tumor archived tissue specimen to test for HLA-G expression.

   In case an archival tissue is not available, patients should be willing to consent for pretreatment biopsy to screen for HLA-G expression.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 [4]
8. Subjects must have adequate venous access for apheresis or agree to use of a central line for apheresis collection.
9. Subject has adequate organ function:

   * Cardiac: Left ventricular ejection fraction (LVEF) at rest must be >45%.
   * Hematologic:

     * Absolute lymphocyte count ≥ 300/μL.
     * Absolute neutrophil count ≥ 1000/μL
     * Platelets ≥ 75,000/μL
     * Hemoglobin ≥ 8.0 g/dL.
   * Hepatic:

     * Total bilirubin ≤ 1.5 x upper limit of normal (ULN), or ≤ 3 x ULN if due to Gilbert's disease
     * Serum aspartate aminotransferase and alanine aminotransferase ≤ 3x ULN, or ≤ 5 x ULN if liver metastases are present.
   * Renal:

     * Creatinine ≤ 1.5 x ULN or eGFR ≥ 50 ml/min
10. From the time of Screening/Study Treatment ICF signature, a female subject must be either:

    * Not of childbearing potential defined as:

      * Postmenopausal (> 45 years of age with amenorrhea ≥ 12 months).
      * Permanently sterilized.
      * Otherwise, incapable of pregnancy.
    * Of childbearing potential and agrees to use 2 highly effective methods of birth control (Effectiveness of Contraception Methods, Centers for Disease Control [CDC] 2018) before lymphodepletion and for at least 12 months after lymphodepletion
11. From the time of Screening/Study Treatment ICF signature, male subjects with female partners of childbearing potential must agree to use 2 highly effective methods of birth control (Effectiveness of Contraception Methods, CDC 2018) for at least 12 months after the last dose of IVS-3001.

Exclusion Criteria:

Subjects who meet any of the following criteria are NOT eligible for the study.

1. Immunotherapy at enrollment and after. Note: Bridging therapies (including herbal therapies) other than immunotherapies are allowed from cell harvest to 2 weeks before lymphodepletion (5 weeks for nitrosoureas or mitomycin) or 5 half-lives, whichever is shorter and must be reported in the CRF.

   Palliative radiotherapy is permitted but treatment must be completed at least 2 weeks prior to the start of lymphodepletion.
2. Symptomatic, untreated, or actively progressing central nervous system metastases (subjects with prior brain metastases treated at least 2 weeks prior to the planned IVS-3001 infusion who are clinically stable and do not require chronic corticosteroid treatment are allowed.
3. Primary CNS tumors.
4. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, or leptomeningeal disease.
5. Ongoing toxicities related to prior anticancer therapy that have not resolved to Grade ≤ 1 (other than alopecia). Note: Current unresolved Grade ≥ 2 non-hematologic toxicity may be allowed after discussing with the study Chair/Co-Chair.
6. Participation in any investigational drug study within 4 weeks prior to cell infusion.
7. Autoimmune disease, chronic infection or any disease requiring systemic immunosuppressive therapy (e.g., calcineurin inhibitors, methotrexate, immunosuppressive antibodies such as anti-IL-6 or anti-IL-6-receptor).
8. Prior CAR T cell or other genetically modified T cell therapy.
9. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   * Symptomatic congestive heart failure requiring treatment.
   * Clinically significant cardiac arrhythmia.
   * Uncontrolled hypertension Acute myocardial infarction or unstable angina pectoris within 6 months prior to enrollment.
   * QTcF > 480 msec; or, marked limitation of physical activity due to symptoms, or unable to carry on any physical activity without discomfort (New York Heart Association Functional Class III-IV).
10. Major surgical procedure, other than for diagnosis, within 4 weeks prior to enrollment, or anticipation of the need for a major surgical procedure during the study.
11. Received a vaccine containing live virus within 6 weeks prior the lymphodepletion.
12. Treatment with systemic chronic steroid therapy (prednisone ≥ 10 mg/day or equivalent) or any other immunosuppressive therapy (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 7 days or 7 half- lives of the prescribed therapy, whichever is shorter, prior to the planned apheresis date.

    Note:
    * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
    * Patients who receive low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
13. Uncontrolled intercurrent illness including but not limited to poorly controlled hypertension or diabetes, or any medical condition determined by the investigator to be a risk for enrolling in the protocol.
14. Untreated or active infection at the time of initial screening, within 72 hours before lymphodepletion or at the time of leukapheresis. Prior oral or IV antibiotics antifungals or antiviral medications must be completed at least 1 week prior to IVS-3001 infusion except for use of prophylactic antimicrobial agents.
15. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of Screening:

    * Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test during Screening. Subjects with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBc Ab) test at screening are eligible for the study if HBV deoxyribonucleic acid (DNA) test is negative. If a subject has a negative HBsAg test and a positive total HBc Ab test at screening, an HBV DNA test should be performed HBV viral load must be less than 100 UI/mL evaluated by PCR
    * Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test during Screening. The HCV RNA test will be performed only for subjects who have a positive HCV test. If patient infected with HBV the viral load must be less than 100 UI/mL evaluated by PCR.
16. History of Grade ≥ 2 bleeding within 4 weeks.
17. Subjects with symptomatic intrinsic lung disease
18. Subject is a woman of child-bearing potential and is pregnant (positive serum β-human choriogonadotropin test at Baseline), planning to become pregnant within 12 months after lymphodepletion, or is breastfeeding.
19. Subject is a man who plans to donate sperm or father a child within 12 months after lymphodepletion.
20. History of second primary malignant disease with the following exceptions:

    * Malignancies that were treated and have not recurred within 2 years prior to Screening.
    * Completely resected basal cell or squamous cell skin cancers.
    * Any malignancy considered to be indolent, not requiring therapy and with low metastatic potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2029-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion an average of 3 years.
. Objective Response Rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | through study completion an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org